CLINICAL TRIAL: NCT04382313
Title: Effect of Hydration Guided by Vigileo on the Prevention of Contrast Induced Nephropathy After Emergency PCI for Patients With Acute Myocardial Infarction
Brief Title: Effect of Hydration Guided by Vigileo on the Prevention of CIN After PCI for Patients With AMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Lu jiang hospital (Unknown)
Responsible Party: Principal Investigator, Qian geng, Clinical Professor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: sf2020-2-5012
Record Dates: First submitted 2020-05-07; First posted 2020-05-11 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-01

CONDITIONS: Myocardial Infarction; Contrast-induced Nephropathy
Keywords: Hydration; Contrast-induced Nephropathy; contrast induced acute kidney injury
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the adequate hydration group guided by Vigileo (Placebo Comparator): The hydration speed is adjusted according to SVV or SV by Vigileo
  Interventions: Procedure: the adequate hydration group guided by Vigileo
- the control group (No Intervention): The routine hydration regimen is adopted, perioperative saline ≤500 ml hydration

INTERVENTIONS:
Procedure: the adequate hydration group guided by Vigileo — If the patient is mechanically ventilated, the following scheme is adopted: if SVV≤10%, then adjust the rehydration speed to 1 ml/kg/h; if 10%<SVV<15%, then adjust the rehydration speed to 2 ml/kg/h; if SVV≥15%, then adjust the rehydration speed to 3 ml/kg/h. The hydration lasts 24 hours after operation, and the rehydration speed is changed according to the SVV. If the patient does not use mechanical ventilation, the following scheme is adopted: 250ml normal saline is administered within 10 minutes after direct PCI, and the rehydration volume changes to 125ml in patients with mild-to-moderate congestive heart failure. If the increment of SV≥15%, then adjust the rehydration speed to 3 ml/kg/h; if 10%≤the increment of SV<15%, then adjust the rehydration speed to 2 ml/kg/h; if the increment of SV<10%, then adjust the rehydration speed to 1 ml/kg/h. Reassessed every 1 hour until SV is stable，and the hydration also lasts 24 hours after operation.
  Arms: the adequate hydration group guided by Vigileo

SUMMARY:
In this study, Vigileo is used to guide hydration adjustment, and SCr is used to estimate renal function. The aim of the study is to investigate the preventive effect of adequate hydration guided by Vigileo on contrast induced nephropathy in patients with acute myocardial infarction who undergo PCI.

DETAILED DESCRIPTION:
This study was conducted in patients with acute myocardial infarction who undergo emergency PCI in Chinese PLA General Hospital. The patients were randomly divided into two groups: the adequate hydration group guided by Vigileo and control group. For the adequate hydration group guided by Vigileo, Vigileo equipment is used to perform hemodynamic monitoring through the femoral or radial arteries to obtain relevant hemodynamic parameters (CO, SV, SVV), and the fluid-rehydration velocity of normal saline is adjusted according to the hemodynamic parameters, and the hydration also lasts 24 hours after operation. For the control group, the routine hydration regimen is adopted, perioperative saline ≤500 ml hydration. The changes of renal function (serum creatinine, serum cystatin), symptoms and signs of cardiac insufficiency during perioperative period and cardiac objective indexes are observed. The incidence of postoperative acute pulmonary edema is recorded, and the major cardiovascular events and hemodialysis events are followed up for 6 months. By comparing the perioperative indexes of heart and kidney function between the intervention group and the control group, the preventive effect of adequate hydration guided by Vigileo on contrast induced nephropathy after PCI was clarified.

ELIGIBILITY:
Inclusion Criteria:

* Clearly diagnosed STEMI or NSTEMI patients:
* Patients aged 18-80 years
* Patients are scheduled to undergo emergency percutaneous coronary interventions
* Estimated glomerular filtration rate eGFR <120ml / min (according to MDRD formula)
* Sign the informed consent to join the group.

Exclusion Criteria:

* Patients with mechanical complications
* Patients with cardiogenic shock
* Patients with aortic dissection
* Patients who have malignant tumors or short-term progressive diseases that researchers believe improper to be included in the group
* Hemodialysis-dependent patients with end-stage renal failure
* Patients who had a history of exposure to radioactive contrast media within 1 week before or 72 hours after direct PCI
* Patients who are allergic to radioactive contrast agents
* Patients diagnosed with right ventricular myocardial infarction with hypotension (defined as systolic blood pressure ≤90 mmHg) on admission.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
Contrast induced nephropathy | 48-72 hours after PCI
  Contrast induced nephropathy is defined as serum creatinine values increased by 0.5 mg/dl or 25% relative to baseline absolute values after direct PCI within 48-72 hours.

SECONDARY OUTCOMES:
The acute renal injury caused by contrast agent | 48 hours after PCI
  The acute renal injury caused by contrast agent is defined as the serum creatinine value increased by 0.3 mg/dl than the baseline absolute value after direct PCI within 48 hours.
Persistent renal insufficiency | 3 months after PCI
  Persistent renal insufficiency is defined as at least 25% decrease compared with baseline in creatinine clearance 3 months after direct PCI.
renal replacement therapy and/or death from acute renal failure | 6 months after PCI
  renal replacement therapy and/or death from acute renal failure
Major adverse cardiac events | 6 months after PCI
  all-cause death, non-lethal acute myocardial infarction, revascularization

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese People's Liberation Army General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Mehran R, Aymong ED, Nikolsky E, Lasic Z, Iakovou I, Fahy M, Mintz GS, Lansky AJ, Moses JW, Stone GW, Leon MB, Dangas G. A simple risk score for prediction of contrast-induced nephropathy after percutaneous coronary intervention: development and initial validation. J Am Coll Cardiol. 2004 Oct 6;44(7):1393-9. doi: 10.1016/j.jacc.2004.06.068. PMID 15464318
- [Background] From AM, Bartholmai BJ, Williams AW, Cha SS, McDonald FS. Mortality associated with nephropathy after radiographic contrast exposure. Mayo Clin Proc. 2008 Oct;83(10):1095-100. doi: 10.4065/83.10.1095. PMID 18828968
- [Background] Sadeghi HM, Stone GW, Grines CL, Mehran R, Dixon SR, Lansky AJ, Fahy M, Cox DA, Garcia E, Tcheng JE, Griffin JJ, Stuckey TD, Turco M, Carroll JD. Impact of renal insufficiency in patients undergoing primary angioplasty for acute myocardial infarction. Circulation. 2003 Dec 2;108(22):2769-75. doi: 10.1161/01.CIR.0000103623.63687.21. Epub 2003 Nov 24. PMID 14638545
- [Background] Marenzi G, Lauri G, Assanelli E, Campodonico J, De Metrio M, Marana I, Grazi M, Veglia F, Bartorelli AL. Contrast-induced nephropathy in patients undergoing primary angioplasty for acute myocardial infarction. J Am Coll Cardiol. 2004 Nov 2;44(9):1780-5. doi: 10.1016/j.jacc.2004.07.043. PMID 15519007
- [Background] Caspi O, Habib M, Cohen Y, Kerner A, Roguin A, Abergel E, Boulos M, Kapeliovich MR, Beyar R, Nikolsky E, Aronson D. Acute Kidney Injury After Primary Angioplasty: Is Contrast-Induced Nephropathy the Culprit? J Am Heart Assoc. 2017 Jun 24;6(6):e005715. doi: 10.1161/JAHA.117.005715. PMID 28647690
- [Background] Pyxaras SA, Sinagra G, Mangiacapra F, Perkan A, Di Serafino L, Vitrella G, Rakar S, De Vroey F, Santangelo S, Salvi A, Toth G, Bartunek J, De Bruyne B, Wijns W, Barbato E. Contrast-induced nephropathy in patients undergoing primary percutaneous coronary intervention without acute left ventricular ejection fraction impairment. Am J Cardiol. 2013 Mar 1;111(5):684-8. doi: 10.1016/j.amjcard.2012.11.018. Epub 2012 Dec 19. PMID 23261003
- [Background] Brar SS, Aharonian V, Mansukhani P, Moore N, Shen AY, Jorgensen M, Dua A, Short L, Kane K. Haemodynamic-guided fluid administration for the prevention of contrast-induced acute kidney injury: the POSEIDON randomised controlled trial. Lancet. 2014 May 24;383(9931):1814-23. doi: 10.1016/S0140-6736(14)60689-9. PMID 24856027
- [Background] Pannu N, Wiebe N, Tonelli M; Alberta Kidney Disease Network. Prophylaxis strategies for contrast-induced nephropathy. JAMA. 2006 Jun 21;295(23):2765-79. doi: 10.1001/jama.295.23.2765. PMID 16788132
- [Background] Task Force on Myocardial Revascularization of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS); European Association for Percutaneous Cardiovascular Interventions (EAPCI); Wijns W, Kolh P, Danchin N, Di Mario C, Falk V, Folliguet T, Garg S, Huber K, James S, Knuuti J, Lopez-Sendon J, Marco J, Menicanti L, Ostojic M, Piepoli MF, Pirlet C, Pomar JL, Reifart N, Ribichini FL, Schalij MJ, Sergeant P, Serruys PW, Silber S, Sousa Uva M, Taggart D. Guidelines on myocardial revascularization. Eur Heart J. 2010 Oct;31(20):2501-55. doi: 10.1093/eurheartj/ehq277. Epub 2010 Aug 29. No abstract available. PMID 20802248
- [Background] Tumkur SM, Vu AT, Li LP, Pierchala L, Prasad PV. Evaluation of intra-renal oxygenation during water diuresis: a time-resolved study using BOLD MRI. Kidney Int. 2006 Jul;70(1):139-43. doi: 10.1038/sj.ki.5000347. Epub 2006 Mar 29. PMID 16572109
- [Background] Epstein FH, Veves A, Prasad PV. Effect of diabetes on renal medullary oxygenation during water diuresis. Diabetes Care. 2002 Mar;25(3):575-8. doi: 10.2337/diacare.25.3.575. PMID 11874950
- [Background] Briguori C, Condorelli G. Hydration in contrast-induced acute kidney injury. Lancet. 2014 May 24;383(9931):1786-8. doi: 10.1016/S0140-6736(14)60753-4. No abstract available. PMID 24856014
- [Background] Bagai A, Armstrong PW, Stebbins A, Mahaffey KW, Hochman JS, Weaver WD, Patel MR, Granger CB, Lopes RD. Prognostic implications of left ventricular end-diastolic pressure during primary percutaneous coronary intervention for ST-segment elevation myocardial infarction: Findings from the Assessment of Pexelizumab in Acute Myocardial Infarction study. Am Heart J. 2013 Nov;166(5):913-9. doi: 10.1016/j.ahj.2013.08.006. Epub 2013 Sep 24. PMID 24176448
- [Background] Remmelink M, Sjauw KD, Henriques JP, Vis MM, van der Schaaf RJ, Koch KT, Tijssen JG, de Winter RJ, Piek JJ, Baan J Jr. Acute left ventricular dynamic effects of primary percutaneous coronary intervention from occlusion to reperfusion. J Am Coll Cardiol. 2009 Apr 28;53(17):1498-502. doi: 10.1016/j.jacc.2008.12.058. PMID 19389559
- [Background] Satiroglu O, Cicek Y, Bostan M, Cetin M, Bozkurt E. Acute change in left ventricle end-diastolic pressure after primary percutaneous coronary intervention in patients with ST segment elevation myocardial infarction. Am Heart Hosp J. 2010 Winter;8(2):E86-90. PMID 21928186
- [Background] Marenzi G, Ferrari C, Marana I, Assanelli E, De Metrio M, Teruzzi G, Veglia F, Fabbiocchi F, Montorsi P, Bartorelli AL. Prevention of contrast nephropathy by furosemide with matched hydration: the MYTHOS (Induced Diuresis With Matched Hydration Compared to Standard Hydration for Contrast Induced Nephropathy Prevention) trial. JACC Cardiovasc Interv. 2012 Jan;5(1):90-7. doi: 10.1016/j.jcin.2011.08.017. PMID 22230154
- [Background] Maioli M, Toso A, Leoncini M, Micheletti C, Bellandi F. Effects of hydration in contrast-induced acute kidney injury after primary angioplasty: a randomized, controlled trial. Circ Cardiovasc Interv. 2011 Oct 1;4(5):456-62. doi: 10.1161/CIRCINTERVENTIONS.111.961391. Epub 2011 Oct 4. PMID 21972403
- [Background] Qian G, Fu Z, Guo J, Cao F, Chen Y. Prevention of Contrast-Induced Nephropathy by Central Venous Pressure-Guided Fluid Administration in Chronic Kidney Disease and Congestive Heart Failure Patients. JACC Cardiovasc Interv. 2016 Jan 11;9(1):89-96. doi: 10.1016/j.jcin.2015.09.026. Epub 2015 Dec 9. PMID 26685074
- [Background] Sugasawa Y, Hayashida M, Yamaguchi K, Kajiyama Y, Inada E. Usefulness of stroke volume index obtained with the FloTrac/ Vigileo system for the prediction of acute kidney injury after radical esophagectomy. Ann Surg Oncol. 2013 Nov;20(12):3992-8. doi: 10.1245/s10434-013-3084-5. PMID 23797754
- [Background] Hofer CK, Senn A, Weibel L, Zollinger A. Assessment of stroke volume variation for prediction of fluid responsiveness using the modified FloTrac and PiCCOplus system. Crit Care. 2008;12(3):R82. doi: 10.1186/cc6933. Epub 2008 Jun 20. PMID 18570641
- [Background] Hofer CK, Muller SM, Furrer L, Klaghofer R, Genoni M, Zollinger A. Stroke volume and pulse pressure variation for prediction of fluid responsiveness in patients undergoing off-pump coronary artery bypass grafting. Chest. 2005 Aug;128(2):848-54. doi: 10.1378/chest.128.2.848. PMID 16100177
- [Background] Sander M, Spies CD, Berger K, Grubitzsch H, Foer A, Kramer M, Carl M, von Heymann C. Prediction of volume response under open-chest conditions during coronary artery bypass surgery. Crit Care. 2007;11(6):R121. doi: 10.1186/cc6181. PMID 18034888
- [Derived] Ling W, Jiang Z, Liu K, Zhang H, Qian Y, Tian J, Zhang Z, Chen Y, Qian G. Effect of Vigileo/FloTrac System-Guided Aggressive Hydration in Acute Myocardial Infarction Patients to Prevent Contrast-Induced Nephropathy After Urgent Percutaneous Coronary Intervention. Am J Cardiol. 2023 May 15;195:77-82. doi: 10.1016/j.amjcard.2023.03.001. Epub 2023 Apr 3. PMID 37018968